CLINICAL TRIAL: NCT03175484
Title: The Influence of the Perceived Workload on Performance During High Fidelity Simulation in Surgical Specialty ( Including Anesthesia) and Nurses
Brief Title: Simulation to Assess Cognitive Workload and Task Load IndeX (TLX) Performance
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, MD, Claude Bernard University
Other Study IDs: HFS-TLX-Lyon
Record Dates: First submitted 2017-05-29; First posted 2017-06-05 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: High Fidelity Simulation; Cognitive Load; Simulation Training/methods*; Task Performance and Analysis*; Students, Medical; Prospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation TLX: surgical specialty ( including anesthesia) residents and nurses undergoing High Fidelity Simulation scenarios.

SUMMARY:
High-fidelity simulation (HFS) is a learning method extensively used for training of surgical specialty (including anesthesia) and nurses. It has a beneficial effect on knowledge of algorithms, team working, early warning scores, and communication. Various skills can be learned using a standardized simulation programs.

The complexity of instructional design may produce cognitive overload, high stress level and anxiety. This may increase fatigue, facilitate errors, and is associated with inferior task performance which may impede memorization of learned skills resulting in inefficient learning/simulation failure. Subjectively reported scales can accurately identify the level of perceived workload and mental demand in individuals during simulation tasks. One example is the National Aeronautics and Space Administration (NASA)-TLX - the most accepted subjective measure of human workload in various industries including medicine.

Surgical specialty (including anesthesia) and nurses training curriculum in Lyon, France, includes several HFS scenarios with a large panel of critical events. The investigators aim to evaluate the effect of burden of workload and stress perceived by surgical specialty (including anesthesia) residents and nurses during HFS on the learning performance, and to grade different learning scenarios by their difficulty.

DETAILED DESCRIPTION:
In this observational study investigators aim to measure anesthesiology, surgeon residents and nurses' workload, stress level, and performance on high-fidelity simulation scenarios used routinely in the current anesthesiology, nurse and surgical training curriculum. A NASA TLX scale, 100 points numeric scale for anxiety (0 - no anxiety; 100 - maximal anxiety), automated quantitative pupillometry, Team Emergency Assessment Measure scale will be used to evaluate a workload, anxiety, stress, and performance. Age, sex, previous experience of HFS will be noted. All data will be anonymized. The participation in this study is voluntary and one can withdraw from this study at any time prior to or after the completion of any interview without any penalty.

Two investigators will independently evaluate the performance of HFS by direct observation and video record if necessary. NASA TLX questionnaire will be administrated immediately after HFS scenario and before the debriefing. Anxiety scale and pupillometry will be administrated before the beginning of HFS scenario and upon its completion.

ELIGIBILITY:
Inclusion Criteria:

* Lyon University medical student status on the day of the study
* Enrolled in surgical specialty (including anesthesia) simulation training program

or

* Lyon Anesthesia Nurses School student status on the day of the study
* Enrolled in surgical specialty (including anesthesia) simulation training program
* voluntary

Exclusion Criteria:

* denial to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All medical students/nurse students enrolled in anesthesia/ surgeon simulation training and participating in the HFS training sessions of June 2017
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Task Load | immediately after the scenario
  NASA TLX scale questionnaire

SECONDARY OUTCOMES:
Anxiety scale | at baseline, at 20 minutes and at 60 minutes
  100 points numeric scale for anxiety (0 - no anxiety; 100 - maximal anxiety)
Pupillometry | at baseline, at 20 minutes and at 60 minutes
  automated quantitative pupillometry
HFS performance | at 20 minutes
  Technical and Team Emergency Assessment Measure scale scores

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lilot, MD, Principal Investigator — CLESS
Locations (1):
- CLESS, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No